Data Analysis for Drug Repurposing for Effective Alzheimer's Medicines – Pentoxifylline vs Cilostazol

NCT05635370

July 7, 2023

## 1. Comparison Details

## a. Intended aim(s)

To evaluate the comparative risk of dementia onset between patients treated with <u>Pentoxifylline versus cilostazol</u> for peripheral artery disease (PAD).

## b. Primary endpoint

Incident dementia (i.e., Alzheimer's disease, vascular dementia, senile, presenile, or unspecified dementia, or dementia in other diseases classified elsewhere).

## 2. Person responsible for implementation

Seanna Vine

# 3. Data Source(s)

Medicare, 2008-2018

# 4. Study Design Diagrams





#### 5. Cohort Identification

#### a. Cohort Summary

This study will employ a new user, active comparator, observational cohort study design comparing <u>Pentoxifylline versus Cilostazol</u>. The patients will be required to have continuous enrollment during the baseline period of 365 days before initiation of study drugs (cohort entry/index date). Follow-up for the outcome (dementia) differs between analyses. Follow-up begins the day after drug initiation (analysis 1, 3, 4); 180 days after drug initiation (analysis 2).

#### b. Key details regarding cohort creation

#### Index date:

Day of initiation of new <u>Pentoxifylline versus Cilostazol</u> use

#### Inclusion criteria for analyses 1, 3, 4:

- Aged ≥ 65 years on the index date
- 365 days enrollment in Medicare Parts A, B, and D with no HMO coverage prior to index date
- No use of <u>Pentoxifylline versus Cilostazol</u>, any time prior to index date (all available lookback approach with a minimum of 365 days)
- No diagnosis of dementia any time prior to and including index date
- No history of nursing home admission recorded in any time prior to and including index date
- At least two claims with peripheral artery disease diagnosis recorded in 365 days prior to index date (ICD-9 or ICD-10 codes)<sup>1</sup>

#### Inclusion criteria for analysis 2:

- Aged ≥ 65 years on the index date
- 365 days enrollment in Medicare Parts A, B, and D with no HMO coverage prior to index date
- No use of <u>Pentoxifylline versus Cilostazol</u>, any time prior to index date (all available lookback approach with a minimum of 365 days)
- No diagnosis of dementia any time prior to and including index date
- No history of nursing home admission recorded in any time prior to and including index date
- At least two claims with peripheral artery disease diagnosis recorded in 365 days prior to index date (ICD-9 or ICD-10 codes)<sup>1</sup>

• 180-day continuous use of Pentoxifylline versus Cilostazol starting on the index date

# c. Flowchart of the study cohort assembly

| | Less Excluded Patients | Remaining Patients |
|---|---|---|
| All patients | | 23,466,175 |
| Did not meet cohort entry criteria | -23,393,311 | 72,864 |
| Excluded due to insufficient enrollment | -45,683 | 27,181 |
| Excluded based on Dementia Exclusion | -6,100 | 21,081 |
| Excluded based on Nursing Home Admission | -4,080 | 17,001 |
| Excluded based on Peripheral artery disease Diagnosis | -4,524 | 12,477 |
| Excluded anyone aged <65 at index | -2,079 | 10,398 |
| Patients in Pentoxifylline group | | 1,701 |
| Patients in Cilostazol group | | 8,697 |
| Final cohort | | 10,398 |

# 6. Variables

# a. Exposure-related variables:

# Study drug:

The study exposure of interest is initiation of Pentoxifylline

Comparator:

Cilostazol

# b. Covariates:

| Demographics | |
|--------------|-----------------------------|
| Age | Region |
| Gender | Calendar year of index date |
| Race | Low income subsidy |

| Dementia risk factors | |
|-------------------------|------------------|
| Diabetes Depression | |
| Obesity | Anxiety |
| Hypertension | Bipolar disorder |
| Coronary artery disease | Schizophrenia |

| Markers for healthy behavior, frailty, healthcare use | |
|---|---|
| Smoking | Number of hospitalizations |
| Mammography | Number of physician office visits |
| Colonoscopy | Number of serum creatinine tests ordered |
| Fecal occult blood test | Composite frailty score |
| Influenza vaccination | Number of C-reactive protein tests ordered |
| Pneumococcal vaccination | Osteoporosis |
| Herpes zoster vaccination | Fractures |
| Bone mineral density test | Falls |
| Number of distinct generic agents | Use of supplemental oxygen |
| Number of emergency room visits | Combined comorbidity score |
| Number of outpatient visits | |

| Comedication use | |
|---|---|
| Lithium Diuretics | |
| Anti-epileptic mood stabilizers | Nitrates |
| Anti-epileptics (other than mood stabilizers) | Lipid lowering drugs |

| Atypical antipsychotics | Non-insulin diabetes medications |
|---|---|
| Benzodiazepines | Insulin |
| Serotonin-norepinephrine reuptake Inhibitors | Antidepressants |
| Selective serotonin reuptake inhibitors | Angiotensin II receptor blockers (ARBs) |
| Tricyclic antidepressants (TCAs) | Angiotensin converting enzyme inhibitors (ACEi) |
| Typical antipsychotics | Calcium channel blockers |
| Anticoagulants | Beta blockers |
| Antiplatelet agents | |

| Comorbid conditions | |
|---|---|
| Atrial fibrillation | Chronic liver disease |
| Coronary artery disease | Asthma |
| Heart failure | Ischemic heart disease |
| Stroke or transient ischemic attack | Chronic obstructive pulmonary disease |
| Peripheral vascular disease | Malignancy |
| Hyperlipidemia | Drug or alcohol abuse or dependence |
| Renal dysfunction Venous thromboembolism | |
| Rheumatoid Arthritis | Hypertension |

| Other PAD treatments and PAD severity indicators | |
|---|---|
| Critical limb ischemia Number of cardiologist visits | |
| Thrombolytic therapy | Number of hospitalizations with PAD |
| (streptokinase, urokinase, alteplase, tissue | |
| plasminogen activator (tPA), pro-urokinase, | |
| reteplase, tenecteplase and Staphylokinase) | |

ICD-9, ICD-10, HCPCS, and NDC codes used to define the covariates listed above are available in Appendix A.

- c. Outcome variables and study follow-up:
- <u>Primary outcome</u>: incident dementia, i.e., Alzheimer's disease, vascular dementia, senile, presenile, or unspecified dementia, or dementia in other diseases classified elsewhere. Outcome will be defined by 1 inpatient

claim or 2 outpatient claims in analysis 1, 2, 3. In analysis 4, the outcome will be defined by 1 inpatient or 1 outpatient claims and 1 prescription claim for a symptomatic treatment [donepezil, galantamine, rivastigmine, and memantine] within 6 months of each other with outcome date assigned to second event in the sequence.

Secondary outcomes: Individual component:
Alzheimer's disease

| Condition | ICD-9 and ICD-10 codes |
|---|---|
| Alzheimer's disease | 331.0*, F00*, G30* |
| Vascular dementia | 290.4*, F01* |
| Senile, presenile, or unspecified dementia | 290.0*, 290.1*. 290.3*, 797*, F03* |
| Dementia in other diseases classified elsewhere | 331.1*, 331.2*, 331.7*, 294.1*, F02* |

For analysis 1,3, and 4 the follow-up will start the day after initiation of <u>Pentoxifylline</u> and <u>Cilostazol</u> and will continue until the earliest date of the following events:

- The first occurrence of the outcome of interest
- · The date of end of continuous registration in the database,
- End of the study period,
- Measured death event occurs,
- The date of drug discontinuation, defined as the date of the last continuous treatment episode of the index drug (<u>Pentoxifylline</u> and <u>Cilostazol</u>) plus a defined grace period (i.e., 90 days after the end of the last prescription's days' supply in main analyses).

For analysis 2, the follow-up will start 180 days after initiation of <u>Pentoxifylline</u> and <u>Cilostazol</u> and will continue until the earliest date of the following events:

- The first occurrence of the outcome of interest, unless otherwise specified for selected outcomes,
- · The date of end of continuous registration in the database,
- · End of the study period,
- · Measured death event occurs,
- Maximum allowed follow-up time (1095 days) reached

#### 7. Propensity score analysis

We will use a propensity-score (PS)²-based approach to account for measured confounding in this study. The PS will be calculated as the predicted probability of initiating the exposure of interest (i.e., the repurposing candidate) versus the reference drug conditional on baseline covariates using multivariable logistic regression constructed separately in each data source. On average, patients with similar PSs have similar distribution of potential confounders used to estimate the PS. Therefore, analyses conditioned on the PS provide effect estimates that are free from measured confounding. For all our analyses, initiators of each exposure of interest will be matched with initiators of the reference exposure based on their PS within each data source.³ Pair matching will be conducted using a nearest-neighbor algorithm, which seeks to minimize the distance between propensity scores in each pair of treated and reference patients,⁴ and a caliper of 0.025 on the natural scale of the PS will be used to ensure similarity between the matched patients.⁵

We report multiple diagnostics for PS analysis in this protocol. First, the PS distributional overlap is provided between two groups before and after matching to ensure comparability of these groups.<sup>6</sup> Next, balance in each individual covariate between two treatment groups is reported using standardized differences.<sup>7</sup>

# 8. Table for covariate balance

| | Crude | | | PS-Matched | | |
|---|---|---|---|---|---|---|
| Variable | Pentoxifylline | Cilostazol | or Diff | Pentoxifylline | Cilostazol | St. |
| | (N = 1,701) | (N = 8,697) | St. Diff | (N = 1,687) | (N = 1,687) | Diff |
| Demographics | | | | | | |
| Age, mean (SD) | 76.2 (7.3) | 75.3 (6.9) | 0.13 | 76.2 (7.2) | 76.3 (7.2) | -0.01 |
| Gender, n (%) | | | | | | |
| Male | 828 (48.7) | 4733 (54.4) | -0.12 | 822 (48.7) | 827 (49) | -0.01 |
| Female | 873 (51.3) | 3964 (45.6) | 0.12 | 865 (51.3) | 860 (51) | 0.01 |
| Race, n (%) | | | | | | |
| White | 1386 (81.5) | 7096 (81.6) | 0.00 | 1377 (81.6) | 1347 (79.8) | 0.05 |
| Black | 156 (9.2) | 935 (10.8) | -0.05 | 156 (9.2) | 176 (10.4) | -0.04 |
| Hispanic | 70 (4.1) | 237 (2.7) | 0.08 | 67 (4) | 65 (3.9) | 0.01 |
| Other | 89 (5.2) | 429 (4.9) | 0.01 | 87 (5.2) | 99 (5.9) | -0.03 |
| Region, n (%) | | | | | | |
| Northeast; n (%) | 274 (16.1) | 1697 (19.5) | -0.09 | 272 (16.1) | 288 (17.1) | -0.03 |
| South; n (%) | 795 (46.7) | 3749 (43.1) | 0.07 | 788 (46.7) | 779 (46.2) | 0.01 |
| Midwest; n (%) | 354 (20.8) | 2069 (23.8) | -0.07 | 353 (20.9) | 337 (20) | 0.02 |
| West; n (%) | 273 (16) | 1171 (13.5) | 0.07 | 269 (15.9) | 279 (16.5) | -0.02 |
| Other; n (%) | 5 (0.3) | 11 (0.1) | 0.04 | 5 (0.3) | 4 (0.2) | 0.01 |
| Calendar year of index date, n (%) | | | | | | |
| 2014 | 444 (26.1) | 2016 (23.2) | 0.07 | 436 (25.8) | 435 (25.8) | 0.00 |
| 2015 | 338 (19.9) | 1908 (21.9) | -0.05 | 336 (19.9) | 310 (18.4) | 0.04 |
| 2016 | 335 (19.7) | 1713 (19.7) | 0.00 | 335 (19.9) | 349 (20.7) | -0.02 |
| 2017 | 303 (17.8) | 1606 (18.5) | -0.02 | 300 (17.8) | 296 (17.5) | 0.01 |

| 2018 | 281 (16.5) | 1454 (16.7) | -0.01 | 280 (16.6) | 297 (17.6) | -0.03 |
|---|---|---|---|---|---|---|
| Low income subsidy, n (%) | 464 (27.3) | 2035 (23.4) | 0.09 | 459 (27.2) | 492 (29.2) | -0.04 |
| Dementia risk factors, n (%) | | | | | | |
| Anxiety | 247 (14.5) | 1090 (12.5) | 0.06 | 245 (14.5) | 236 (14) | 0.02 |
| Bipolar disorder | 15 (0.9) | 67 (0.8) | 0.01 | 15 (0.9) | 13 (0.8) | 0.01 |
| Coronary artery disease | 800 (47) | 4789 (55.1) | -0.16 | 792 (46.9) | 790 (46.8) | 0.00 |
| Depression | 240 (14.1) | 1027 (11.8) | 0.07 | 236 (14) | 226 (13.4) | 0.02 |
| Diabetes | 826 (48.6) | 4211 (48.4) | 0.00 | 819 (48.5) | 852 (50.5) | -0.04 |
| Hypertension | 1512 (88.9) | 8055 (92.6) | -0.13 | 1500 (88.9) | 1502 (89) | 0.00 |
| Obesity | 325 (19.1) | 1373 (15.8) | 0.09 | 321 (19) | 308 (18.3) | 0.02 |
| Schizophrenia | 2 (0.1) | 8 (0.1) | 0.01 | | | 0.00 |
| Markers for healthy behavior, frailty, healthcare use | | | | | | |
| Bone mineral density test, n (%) | 141 (8.3) | 725 (8.3) | 0.00 | 139 (8.2) | 130 (7.7) | 0.02 |
| Colonoscopy, n (%) | 143 (8.4) | 861 (9.9) | -0.05 | 141 (8.4) | 148 (8.8) | -0.02 |
| Fecal occult blood test, n (%) | 132 (7.8) | 696 (8) | -0.01 | 131 (7.8) | 131 (7.8) | 0.00 |
| Influenza vaccination, n (%) | 1035 (60.8) | 5419 (62.3) | -0.03 | 1026 (60.8) | 978 (58) | 0.06 |
| Mammography, n (%) | 281 (16.5) | 1455 (16.7) | -0.01 | 279 (16.5) | 283 (16.8) | -0.01 |
| Pneumococcal vaccination, n (%) | 652 (38.3) | 3612 (41.5) | -0.07 | 649 (38.5) | 621 (36.8) | 0.03 |
| Smoking, n (%) | 599 (35.2) | 3881 (44.6) | -0.19 | 595 (35.3) | 580 (34.4) | 0.02 |
| Number of C-reactive protein tests ordered, mean (SD) | 0.3 (1.2) | 0.2 (0.7) | 0.13 | 0.3 (0.9) | 0.3 (1) | -0.02 |
| Number of emergency room visits, mean (SD) | 0.8 (1.4) | 0.7 (1.3) | 0.08 | 0.7 (1.4) | 0.7 (1.4) | 0.00 |
| Number of distinct prescriptions, mean (SD) | 13.9 (6.7) | 12.4 (5.9) | 0.23 | 13.7 (6.6) | 13.8 (6.7) | 0.00 |

# DREAM study protocol - Comparison 12 Pentoxifylline vs Cilostazol

| Number of hospitalizations, mean (SD) | 0.3 (0.7) | 0.2 (0.6) | 0.09 | 0.3 (0.7) | 0.3 (0.6) | 0.01 |
|---|---|---|---|---|---|---|
| Number of outpatient visits, mean (SD) | 15 (10.6) | 13.1 (8.6) | 0.20 | 14.8 (10.1) | 14.9 (10) | -0.01 |
| Number of serum creatinine tests ordered, mean (SD) | 1.6 (2.7) | 1.5 (2.3) | 0.01 | 1.6 (2.7) | 1.5 (2.2) | 0.02 |
| Composite frailty score, mean (SD) | 0.2 (0.1) | 0.2 (0.1) | 0.21 | 0.2 (0.1) | 0.2 (0.1) | 0.02 |
| Falls, n (%) | 107 (6.3) | 472 (5.4) | 0.04 | 107 (6.3) | 108 (6.4) | 0.00 |
| Fractures, n (%) | 141 (8.3) | 591 (6.8) | 0.06 | 139 (8.2) | 138 (8.2) | 0.00 |
| Osteoporosis, n (%) | 247 (14.5) | 1051 (12.1) | 0.07 | 242 (14.3) | 239 (14.2) | 0.01 |
| Use of supplemental oxygen, n (%) | 26 (1.5) | 150 (1.7) | -0.02 | 26 (1.5) | 23 (1.4) | 0.02 |
| Combined comorbidity score, mean (SD) | 3.4 (2.8) | 2.9 (2.4) | 0.18 | 3.3 (2.7) | 3.4 (2.6) | -0.02 |
| Comedication use, n (%) | | | | | | |
| Angiotensin converting enzyme inhibitors (ACEi) | 646 (38) | 3657 (42) | -0.08 | 643 (38.1) | 641 (38) | 0.00 |
| Angiotensin II receptor blockers (ARBs) | 488 (28.7) | 2519 (29) | -0.01 | 485 (28.7) | 482 (28.6) | 0.00 |
| Antidepressants | 435 (25.6) | 2046 (23.5) | 0.05 | 430 (25.5) | 416 (24.7) | 0.02 |
| Beta blockers | 894 (52.6) | 4801 (55.2) | -0.05 | 887 (52.6) | 884 (52.4) | 0.00 |
| Calcium channel blockers | 593 (34.9) | 3243 (37.3) | -0.05 | 588 (34.9) | 590 (35) | 0.00 |
| DMARD | 86 (5.1) | 212 (2.4) | 0.14 | 80 (4.7) | 81 (4.8) | 0.00 |
| Diuretics | 930 (54.7) | 4251 (48.9) | 0.12 | 918 (54.4) | 925 (54.8) | -0.01 |
| Insulin | 228 (13.4) | 1176 (13.5) | 0.00 | 224 (13.3) | 216 (12.8) | 0.01 |
| Lipid lowering drugs | 1169 (68.7) | 6557 (75.4) | -0.15 | 1161 (68.8) | 1151 (68.2) | 0.01 |
| Nitrates | 239 (14.1) | 1355 (15.6) | -0.04 | 233 (13.8) | 225 (13.3) | 0.01 |

# DREAM study protocol - Comparison 12 Pentoxifylline vs Cilostazol

| Non-insulin diabetes medications | 477 (28) | 2493 (28.7) | -0.01 | 473 (28) | 481 (28.5) | -0.01 |
|---|---|---|---|---|---|---|
| Anticoagulants | 218 (12.8) | 814 (9.4) | 0.11 | 212 (12.6) | 190 (11.3) | 0.04 |
| Anti-epileptic mood stabilizers | 20 (1.2) | 94 (1.1) | 0.01 | 20 (1.2) | 17 (1) | 0.02 |
| Antiplatelet agents | 411 (24.2) | 8697 (100) | -2.51 | | | 0.00 |
| Atypical antipsychotics | 25 (1.5) | 102 (1.2) | 0.03 | 25 (1.5) | 22 (1.3) | 0.02 |
| Benzodiazepines | 352 (20.7) | 1416 (16.3) | 0.11 | 347 (20.6) | 331 (19.6) | 0.02 |
| Lithium | 2 (0.1) | 14 (0.2) | -0.01 | | | 0.00 |
| Anti-epileptics (other than mood stabilizers) | 459 (27) | 2073 (23.8) | 0.07 | 455 (27) | 457 (27.1) | 0.00 |
| Serotonin-norepinephrine reuptake inhibitors | 83 (4.9) | 361 (4.2) | 0.04 | 82 (4.9) | 75 (4.4) | 0.02 |
| Selective serotonin reuptake inhibitors | 222 (13.1) | 1141 (13.1) | 0.00 | 221 (13.1) | 221 (13.1) | 0.00 |
| Tricyclic antidepressants (TCAs) | 77 (4.5) | 320 (3.7) | 0.04 | 75 (4.4) | 63 (3.7) | 0.04 |
| Typical antipsychotics | 8 (0.5) | 20 (0.2) | 0.04 | 8 (0.5) | 10 (0.6) | -0.02 |
| Other PAD treatments and PAD severity indicators , n (%) | | | | | | |
| Critical limb ischemia | 394 (23.2) | 1058 (12.2) | 0.29 | 381 (22.6) | 380 (22.5) | 0.00 |
| Thrombolytic therapy | 10 (0.6) | 26 (0.3) | 0.04 | 9 (0.5) | 6 (0.4) | 0.03 |
| Number of cardiologist visits, mean (SD) | 3.5 (5.9) | 4 (5.2) | -0.08 | 3.5 (5.9) | 3.5 (4.9) | -0.01 |
| Number of hospitalizations with PAD, mean (SD) | 0 (0.1) | 0 (0.2) | -0.04 | 0 (0.1) | 0 (0.1) | 0.01 |
| Comorbid conditions, n (%) | | | | | | |
| Atrial fibrillation | 296 (17.4) | 1195 (13.7) | 0.10 | 290 (17.2) | 296 (17.5) | -0.01 |

## DREAM study protocol - Comparison 12 Pentoxifylline vs Cilostazol

| Chronic obstructive pulmonary disease | 557 (32.7) | 2821 (32.4) | 0.01 | 550 (32.6) | 556 (33) | -0.01 |
|---|---|---|---|---|---|---|
| Chronic liver disease | 91 (5.3) | 591 (6.8) | -0.06 | 89 (5.3) | 89 (5.3) | 0.00 |
| Drug or alcohol abuse or dependence | 282 (16.6) | 2134 (24.5) | -0.20 | 281 (16.7) | 284 (16.8) | -0.01 |
| Heart failure | 336 (19.8) | 1320 (15.2) | 0.12 | 329 (19.5) | 335 (19.9) | -0.01 |
| Hyperlipidemia | 1309 (77) | 7176 (82.5) | -0.14 | 1300 (77.1) | 1303 (77.2) | 0.00 |
| Ischemic heart disease | 792 (46.6) | 4714 (54.2) | -0.15 | 784 (46.5) | 783 (46.4) | 0.00 |
| Malignancy | 508 (29.9) | 2426 (27.9) | 0.04 | 502 (29.8) | 517 (30.6) | -0.02 |
| Peripheral vascular disease | 1646 (96.8) | 8451 (97.2) | -0.02 | 1634 (96.9) | 1635 (96.9) | 0.00 |
| Rheumatoid Arthritis | 112 (6.6) | 348 (4) | 0.12 | 108 (6.4) | 100 (5.9) | 0.02 |
| Renal dysfunction | 478 (28.1) | 2178 (25) | 0.07 | 471 (27.9) | 478 (28.3) | -0.01 |
| Stroke or transient ischemic attack | 241 (14.2) | 1170 (13.5) | 0.02 | 236 (14) | 242 (14.3) | -0.01 |
| Venous thromboembolism | 132 (7.8) | 410 (4.7) | 0.13 | 128 (7.6) | 125 (7.4) | 0.01 |

#### 9. Statistical analysis plans

Incidence rates for the outcome will be estimated for the treatment and reference groups before and after PS matching. The competing risk of death could be of concern for the current set of analyses if mortality is frequent among patients included in the cohort and if differences in the risk of mortality between treatment and reference groups are substantial. In the PS-matched sample, we will use cause-specific hazard models<sup>8</sup> to provide hazard ratios averaged over the entire follow-up period as well as interval specific hazard ratios (1, 2, and 3 years) for the association between the treatment of interest and risk of ADRD after considering all-cause mortality as a competing event. Pre-specified subgroup analyses will be conducted based on age, sex, and baseline cardiovascular disease.

#### 10. References

- Weissler EH, Lippmann SJ, Smerek MM, et al. Model-Based Algorithms for Detecting Peripheral Artery Disease Using Administrative Data From an Electronic Health Record Data System: Algorithm Development Study. *JMIR Med Inform*. 2020;8(8):e18542.
- 2. Rosenbaum PR, Rubin DB. The central role of the propensity score in observational studies for causal effects. *Biometrika*. 1983;70(1):41-55.
- Rassen JA, Avorn J, Schneeweiss S. Multivariate-adjusted pharmacoepidemiologic analyses of confidential information pooled from multiple health care utilization databases. *Pharmacoepidemiology and drug safety*. 2010;19(8):848-857.
- 4. Rassen JA, Shelat AA, Myers J, Glynn RJ, Rothman KJ, Schneeweiss S. One-to-many propensity score matching in cohort studies. *Pharmacoepidemiol Drug Saf.* 2012;21 Suppl 2:69-80.
- 5. Austin PC. Some Methods of Propensity-Score Matching had Superior Performance to Others: Results of an Empirical Investigation and Monte Carlo simulations. *Biometrical Journal*. 2009;51(1):171-184.
- 6. AM Walker AM, Patrick A, Lauer M, et al. Tool for Assessing the Feasibility of Comparative Effectiveness Research. *Comp Effect Res* 2013;3:11-20.
- 7. Franklin JM, Rassen JA, Ackermann D, Bartels DB, Schneeweiss S. Metrics for covariate balance in cohort studies of causal effects. *Statistics in medicine*. 2014;33(10):1685-1699.
- 8. Austin PC, Lee DS, Fine JP. Introduction to the analysis of survival data in the presence of competing risks. *Circulation*. 2016;133(6):601-609.